CLINICAL TRIAL: NCT07113548
Title: PERSONAE: a Personalized Adaptation of Stepped Care Internet-based Cognitive Behavioral Therapy for Depression - A Randomized Controlled Trial
Brief Title: PERSONAE - a Personalized Online Treatment of Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Kim Mathiasen, Associate professor, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIV-25-01-050494; 2077-00009B (Other Grant/Funding Number: Innovation Fund Denmark)
Record Dates: First submitted 2025-06-12; First posted 2025-08-08 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Depression - Major Depressive Disorder
Keywords: Depression; iCBT; randomized controlled trial; personalized; stepped-care; internet-based
MeSH Terms: conditions — Depression

STUDY DESIGN:
Masking Description: Since the two conditions are easily distinguishable, care providers and participants will remain blinded until the participant has completed the baseline questionnaires and has been randomized. After randomization, unblinding is unavoidable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PERSONAE (Experimental): Personalized treatment arm
  Interventions: Behavioral: Personalized iCBT for depression
- Treatment As Usual (Active Comparator): Standard iCBT
  Interventions: Behavioral: Standard iCBT

INTERVENTIONS:
Behavioral: Personalized iCBT for depression — Participants receive 12 sessions of personalized treatment in an online iCBT program. The treatment includes the option for weekly written feedback from a psychologist, or video-based interventions depending on the participant's current status. The content of the 12-week program is tailored to the participant's individual symptom profile.
  The treatment incorporates elements from standard Cognitive Behavioral Therapy (CBT), Acceptance and Commitment Therapy (ACT), Compassion-Focused Therapy (CFT), and Positive Activity Interventions (PAT).
  The program consists of nine modules, each targeting a specific area:
  Rumination,
  Anhedonia,
  Tearfulness and emotional regulation,
  Sleep problems,
  Difficulty concentrating,
  Eating issues,
  Low energy,
  Social withdrawal,
  Self-critical thinking,
  The treatment concludes with support aimed at preventing relapse.
  Arms: PERSONAE
Behavioral: Standard iCBT — Standard iCBT consisting of a "one size fits all"" progression of cognitive behavioral therapy over 12 weeks. This includes:
  Introduction to Online Cognitive Behavioral Therapy
  Start of Treatment
  Rumination
  Activity Monitoring
  Activity Planning
  Cognitive Restructuring
  Behavioral Experiment I
  Behavioral Experiment II
  Core Beliefs I
  Core Beliefs II
  Relapse Prevention
  Arms: Treatment As Usual

SUMMARY:
The goal of this clinical trial is to determine whether a personalized online treatment for depression, delivered via an app (PERSONAE), is effective in treating mild to moderate depression in adults. The study will also assess the safety of the Monsenso app. The main questions it aims to answer are:

Does the PERSONAE intervention reduce depression scores compared to standard internet-based treatment for depression?

What challenges do participants experience when using the PERSONAE intervention?

Researchers will compare PERSONAE to Treatment As Usual (a standard, one-size-fits-all treatment) to evaluate whether PERSONAE is more effective in treating mild to moderate depression.

Participants will:

Complete a 12-week online treatment program based on cognitive behavioral therapy (CBT).

Undergo an intake assessment and complete weekly questionnaires.

Receive guidance from a clinical psychologist tailored to their individual needs

DETAILED DESCRIPTION:
Prevalence and cost of depression

Depression is a highly prevalent disorder in Europe (Alonso et al., 2004). Globally, 280 million are estimated to suffer from depression. In Denmark, 13.2% of the population suffers from depression. The cost of affective disorders in Europe was estimated to be 106 billion euros in 2004. In Denmark, the health board's newest estimates of the cost of depression are 6700 deaths a year, 10 billion DKK for treatment, and 25 billion DKK in lost productivity. Depression has been found to cause 1124 quality-adjusted life years (QALY) lost per 100,000 patients, and compared with the general population, patients with mental disorders experience one standard deviation of lower quality of life.

Although depression is highly prevalent both in Denmark and internationally, not enough individuals with depression receive the help they need. There are barriers that can discourage help-seeking behavior. Some of the most important barriers to help-seeking behavior in Denmark are the high costs of psychotherapy as the service costs the patient pays 40% of the costs of the consultations, even after referral, and long waiting lists for being seen at a private practice psychologist. The stigma associated with mental illness, limited number of trained clinicians, and limited access to low-threshold, low-cost, and evidence-based psychotherapy furthermore present significant barriers. Several researchers have recommended further study of the implementation and dissemination of evidence-based psychotherapies.

Cognitive behavioral therapy

Cognitive behavioral therapy - one of the most used and evidence-based forms of therapy - is a combination of behavioral and cognitive therapy. Behavioral therapy was developed in the 1930's and -40's based on the research by e.g. Skinner, Pavlov, and Watson. The underlying assumption is that the patient repeats conditioned dysfunctional behaviors, which can become extinct or counteracted by behavioral exercises e.g. behavioral activation. Cognitive therapy was originally developed by Aaron Beck and is based on observations of occurrences of cognitive distortions or thought patterns that are not realistic or verifiable, leading to the conclusion that thoughts are the cause of depression. Maladaptive assumptions (thoughts) result in maladaptive behavior strategies and the development of maintenance behavior. According to Beck, cognitive distortions are a common trait in all mental disorders, and the treatment should therefore target distortions, thereby enabling awareness and realistic appraisals.

Today, behavioral and cognitive methods are combined and referred to as Cognitive Behavioral Therapy (CBT), which is often denoted second wave CBT. CBT employs both behavioral interventions and working with cognitive distortions.

CBT has been shown to be a clinically- and cost-effective treatment for depression. CBT demonstrates results equal to antidepressant pharmacotherapy and compared with pharmacotherapy only has a longer lasting effect and higher acceptability.

However, CBT still has some shortcomings, such as lack of focus on contextual influences on the patient, lack of focus on accepting negative thoughts that are not distorted, and lack of focus on emotions and emotion regulation. These shortcomings have given rise to a third wave of CBT.

This third-wave CBT consists of several different approaches, each of which tries to cover some of the lack in second-wave CBT. For example, another approach is Acceptance and Commitment Therapy (ACT), which contextualizes a person's situation, and instead of focusing only on distorted thoughts, the focus on acceptance and diffusion from thoughts and emotion is heightened compared to core CBT. Compassion focused therapy (CFT) is based on an evolutionary framework assuming humans are social beings with pro-social behavior that evolved to enhance in-group cohesion. CFT focuses on enhancing the innate compassionate and altruistic abilities towards the depressed person themselves. The purpose is to overcome the base fear and threat modes such as the inner critical voice. CFT as a tool in depression treatment is focused on shame and guilt and can especially aid people who have had adverse childhoods or other shame-inducing experiences. Positive Affect Treatment (PAT) is designed to address the symptom of anhedonia common in depression. Traditional therapies primarily focus on reducing negative emotions, whereas PAT directly targets deficits in the brain's reward system.

Internet-based self-guided, guided, and blended cognitive behavioral therapy

Over the course of the past two decades, researchers have investigated the possibility of delivering CBT via the internet in a guided self-help format named Internet-based Cognitive Behavioral Therapy (iCBT). The main part of the therapy is delivered in a self-help format through an internet-based computer program. These programs use the same therapeutic interventions, as face-to-face therapy formats; however, the content is adapted for delivery via a web platform largely designed to function as self-help. Since iCBT is still based on evidence-based CBT methods, it is not a new treatment in the classical sense, but rather a different treatment delivery format. The temporal structure also largely mimics face-to-face therapy, so patients typically go through one module in the program per week, after which they are given homework assignments, which they are expected to work on for about a week. Hereafter, they log back into the program again and take the next module, and so on. These programs typically contain 6-10 modules typically taken over approximately three months. However, there is great variation in how many modules are taken. The content of the modules are psychoeducation and exercises delivered via a variety of multimedia elements, e.g. video- and audio clips, text passages, graphics, animations, etc. Several meta-analyses have shown this treatment format to be efficacious for depression - particularly when the patients are assessed for eligibility prior to engaging with the programs and are supported by a clinician with even a minimal level of support. The support is usually comprised of approximately 10-20 minutes per week via either telephone or a secure email-like text medium built into the digital platform delivering the treatment content.

However, guided iCBT only targets a specific group of depressed patients. People with low or high symptom severity may be excluded from treatment as well as conditions with complications such as comorbidities (e.g. anxiety) or social problems interfering with the therapy. To embrace a larger demographic, earlier or stabilizing interventions or the possibility of more contact with a clinician should target these demographics. This can be achieved by including two additional treatment delivery formats: self-guided iCBT (S-iCBT) and blended iCBT (B-iCBT).

Self-guided denotes the fact that there is no actual clinician contact, and the main therapeutic alliance is formed with the program itself. There can be technical support, phone support with non-clinical staff, or no support at all. S-iCBT is effective in treating sub-threshold and mild depression. Moreover, S-iCBT has been demonstrated to be less harmful than a waitlist condition, indicating that self-guided programs are safer than no treatment. This is an important point considering that many patients are currently untreated, and a this unmet need could potentially be addressed by a cost-efficient and low-barrier service, such as self-guidet iCBT.

Patients suffering from more severe depression or comorbid disorders may need more clinician contact and support. This is especially true of those at risk of dropping out of treatment. In these cases, blended care iCBT (B-iCBT) can be employed. This type of iCBT consists of a mix of video/face-to-face consultations with a clinician and online exercises in a digital program. This format was tested in a randomized study on the clinical effectiveness of B-iCBT and was compared to face-to-face CBT for depression. In this study, it was found that although the blended condition only received half the consultations as the face-to-face condition, attrition rates and effects of treatment were similar in the two conditions. In a large-scale EU study, e-Compared, the effectiveness of B-iCBT was comparable to or better than face-to-face treatment. These two studies indicate effectiveness of B-CBT, in a patient population with moderate to severe symptom levels compared to treatment as usual in primary and secondary care.

The heterogeneous nature of depression

Symptoms of depression include rumination, guilt and shame, sleep problems, depressed mood, anhedonia, concentration difficulties, low energy/fatigue, agitation/inhibition, weight changes and suicidal ideations.

Per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) there are 256 different combinations of symptoms that will lead to a diagnosis of depression, some of which are opposites (sleeping too much or too little or gaining or losing weight). Unipolar depression can be further divided into subtypes such as melancholic, seasonal, anxious, psychotic or atypical and they have varying characteristics such as onset, severity and recurrence. The same person can also experience different types of depression across a lifespan. Based on this heterogeneous nature, personalized treatment for depression is warranted. The problem is that iCBT for depression as it has been offered until now, is a very inflexible treatment that is often delivered as a "one-size-fits-all" approach to therapy. One approach to overcome this problem with iCBT is to engage in a care model, which adapts to the patient's needs regarding treatment intensity (self-guided, guided, or blended care) and to personalize the content based on each person's manifestation of depression.

Drop-out rates and predictors of adherence

Drop-out rates in iCBT vary widely in different conditions. A meta-analysis from 2012 found that in a completely self-guided setting, the drop-out rate was 74%. With administrative support, the drop-out rate decreased to 38%, and with non-clinical staff supporting treatment, it decreased to 28%. In a meta-analysis from Karyotaki et al., 2015, predictors for drop-out in guided iCBT were found to be male gender, lower educational level, and younger age. Furthermore, patients reported that drop-out could be caused by interference from external parameters that exist apart from the treatment itself, e.g., relationship problems and work scheduling issues, or from internal factors such as dissatisfaction with treatment allocation, time constrains, lack of treatment effect, not understanding how the programs work, or technical issues. Interestingly, some patients dropout because their condition improves. Higher rates of drop-out have also been found in people low in neuroticism and high in openness to experience. Conversely, extroversion and patients' ability to acquire new skills has been associated with completion. Importantly, it has been found that patients are more likely to stay committed to treatment if the treatment is experienced as meaningful for them and fosters motivation.

Dose dependent effect

Earlier evidence from traditional psychotherapy suggests that 11-13 sessions are needed for participants to have received adequate treatment and attain an effect on mental health problems. In the newer literature discussing iCBT and the effectiveness of CBT in general, an adequate dose is used to describe the saturation where participants have received enough treatment for it to work and last. The dose is often designated as 75% of the planned treatment or eight sessions.

Motivation for treatment

When learning new skills, such as when children start learning mathematics or languages, it is generally assumed that starting with small steps is the best approach. Children start learning at a simple level and move up in complexity by staying in the zone of proximal development. The zone of proximal development was defined by Vygotsky as the next step for learning new skills, with the help from adults or, more relevant for psychotherapy, more capable peers. This stepwise rise in complexity grants you experiences of success, which, in turn, fosters intrinsic motivation. Today this method has been augmented and is better known as scaffolding. Psychotherapy, especially CBT, can be compared to learning new skills as a clinician enables patients to understand and change dysfunctional learned and innate behavior through the patients' process of change and identification. Therefore, if depression treatment is scaled based on the level the participant is currently able to understand and profit from, it could provide more experiences of success and enable more autonomy, relatedness and experience of competency.

To increase adherence and effect of the treatment, the treatment has been developed to be meaningful for the individual patient, to target heterogenuity of depression and designed to be self-guidet, guidet and blended depending on the individual need of participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Patient Health Questionnaire-9 items (PHQ-9) >4 AND <22.
* Any gender.
* Meeting the diagnostic criteria of the International Classification of Diseases and Related Health Problems 10th edition for major depressive disorder

Exclusion Criteria:

* Unable to speak and/or read Danish.
* No access to a smartphone.
* Pregnant or breastfeeding.
* Heightened suicide risk as per the PHQ-9 (item 9 >1) and Quick Inventory of Depressive Symptoms (QIDS) item 12.
* Comorbid disorders: Diagnosed substance dependence, bipolar affective disorder, psychotic illness, or obsessive-compulsive disorder.
* Not currently in therapeutic treatment for anxiety or depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the mean depression score on the 9-item Patient Health Questionnaire (PHQ-9). | From enrollment to 12 weeks of treatment, plus follow up at 3, 6, and 12 months
  The Patient Health Questionnaire-9 (PHQ-9) has a total score range of 0-27, with higher scores indicating more severe depressive symptoms. The questionnaire will be administered via automated REDCap surveys at baseline, post-treatment, and at 3-, 6-, and 12-month follow-ups, as well as during treatment through the Minddistrict (TAU) and Monsenso (PERSONAE) programs. The PHQ-9 evaluates nine core symptoms of depression.

SECONDARY OUTCOMES:
Adherence rates | This will be assessed at the individual patient level, once the patient is no longer active in treatment-either due to completing the 12-week program or discontinuing active engagement with the intervention.
  Adherence will be measured as a binary outcome, defined by whether participants have completed at least 75% of the designated treatment content or have been active for at least 75% of the allotted treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Mathiasen, Ph.d., Principal Investigator — University of Southern Denmark & Aarhus University
Locations (1):
- Center for Digital Psychiatry, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
After the study period, de-identified data will be shared with the University of Limerick to support the development of an algorithm aimed at helping clinicians identify at-risk patients, determine appropriate treatment content, and enhance screening efforts.
Supporting Information: Study Protocol, SAP
Time Frame: Q3 2025 to Q2 2027
Access Criteria: Pepijn van de Ven is a Professor in the Department of Electronic and Computer Engineering at the University of Limerick. Data will be shared via Jupyter. A data use agreement has been approved, and each participant provides separate consent for data sharing. If a participant declines, their data will be excluded prior to sharing.

REFERENCES:
- [Background] Videbech P, Deleuran A. The Danish Depression Database. Clin Epidemiol. 2016 Oct 25;8:475-478. doi: 10.2147/CLEP.S100298. eCollection 2016. PMID 27843341
- [Background] Andersson G, Bergstrom J, Hollandare F, Carlbring P, Kaldo V, Ekselius L. Internet-based self-help for depression: randomised controlled trial. Br J Psychiatry. 2005 Nov;187:456-61. doi: 10.1192/bjp.187.5.456. PMID 16260822
- [Background] Andrews G, Cuijpers P, Craske MG, McEvoy P, Titov N. Computer therapy for the anxiety and depressive disorders is effective, acceptable and practical health care: a meta-analysis. PLoS One. 2010 Oct 13;5(10):e13196. doi: 10.1371/journal.pone.0013196. PMID 20967242
- [Background] Barney LJ, Griffiths KM, Jorm AF, Christensen H. Stigma about depression and its impact on help-seeking intentions. Aust N Z J Psychiatry. 2006 Jan;40(1):51-4. doi: 10.1080/j.1440-1614.2006.01741.x. PMID 16403038
- [Background] Brown LA, Gaudiano BA, Miller IW. Investigating the similarities and differences between practitioners of second- and third-wave cognitive-behavioral therapies. Behav Modif. 2011 Mar;35(2):187-200. doi: 10.1177/0145445510393730. PMID 21324946
- [Background] Buch AM, Liston C. Dissecting diagnostic heterogeneity in depression by integrating neuroimaging and genetics. Neuropsychopharmacology. 2021 Jan;46(1):156-175. doi: 10.1038/s41386-020-00789-3. Epub 2020 Aug 11. PMID 32781460
- [Background] Carlbring P, Andersson G, Cuijpers P, Riper H, Hedman-Lagerlof E. Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: an updated systematic review and meta-analysis. Cogn Behav Ther. 2018 Jan;47(1):1-18. doi: 10.1080/16506073.2017.1401115. Epub 2017 Dec 7. PMID 29215315
- [Background] Cuijpers P, Reijnders M, Karyotaki E, de Wit L, Ebert DD. Negative effects of psychotherapies for adult depression: A meta-analysis of deterioration rates. J Affect Disord. 2018 Oct 15;239:138-145. doi: 10.1016/j.jad.2018.05.050. Epub 2018 Jul 3. PMID 30005327
- [Background] Donkin L, Glozier N. Motivators and motivations to persist with online psychological interventions: a qualitative study of treatment completers. J Med Internet Res. 2012 Jun 22;14(3):e91. doi: 10.2196/jmir.2100. PMID 22743581
- [Background] Etzelmueller A, Vis C, Karyotaki E, Baumeister H, Titov N, Berking M, Cuijpers P, Riper H, Ebert DD. Effects of Internet-Based Cognitive Behavioral Therapy in Routine Care for Adults in Treatment for Depression and Anxiety: Systematic Review and Meta-Analysis. J Med Internet Res. 2020 Aug 31;22(8):e18100. doi: 10.2196/18100. PMID 32865497
- [Background] Folker AP, Mathiasen K, Lauridsen SM, Stenderup E, Dozeman E, Folker MP. Implementing internet-delivered cognitive behavior therapy for common mental health disorders: A comparative case study of implementation challenges perceived by therapists and managers in five European internet services. Internet Interv. 2018 Feb 6;11:60-70. doi: 10.1016/j.invent.2018.02.001. eCollection 2018 Mar. PMID 30135761
- [Background] Goldberg D. The heterogeneity of "major depression". World Psychiatry. 2011 Oct;10(3):226-8. doi: 10.1002/j.2051-5545.2011.tb00061.x. No abstract available. PMID 21991283
- [Background] Grandes G, Montoya I, Arietaleanizbeaskoa MS, Arce V, Sanchez A; MAS Group. The burden of mental disorders in primary care. Eur Psychiatry. 2011 Oct;26(7):428-35. doi: 10.1016/j.eurpsy.2010.11.002. Epub 2011 Feb 8. PMID 21306876
- [Background] Gunter RW, Whittal ML. Dissemination of cognitive-behavioral treatments for anxiety disorders: Overcoming barriers and improving patient access. Clin Psychol Rev. 2010 Mar;30(2):194-202. doi: 10.1016/j.cpr.2009.11.001. Epub 2009 Nov 10. PMID 19942331
- [Background] Gustavsson A, Svensson M, Jacobi F, Allgulander C, Alonso J, Beghi E, Dodel R, Ekman M, Faravelli C, Fratiglioni L, Gannon B, Jones DH, Jennum P, Jordanova A, Jonsson L, Karampampa K, Knapp M, Kobelt G, Kurth T, Lieb R, Linde M, Ljungcrantz C, Maercker A, Melin B, Moscarelli M, Musayev A, Norwood F, Preisig M, Pugliatti M, Rehm J, Salvador-Carulla L, Schlehofer B, Simon R, Steinhausen HC, Stovner LJ, Vallat JM, Van den Bergh P, van Os J, Vos P, Xu W, Wittchen HU, Jonsson B, Olesen J; CDBE2010Study Group. Cost of disorders of the brain in Europe 2010. Eur Neuropsychopharmacol. 2011 Oct;21(10):718-79. doi: 10.1016/j.euroneuro.2011.08.008. Epub 2011 Sep 15. PMID 21924589
- [Background] Isabelle Mairey, S. R., Marie Borring Klitgaard og Lau Caspar Thygesen,. (2022). Sygdomsbyrden i Danmark - sygdomme. København: Sundhedsstyrelsen Islands Brygge 67 2300 København S
- [Background] Mathiasen K, Riper H, Andersen TE, Roessler KK. Guided Internet-Based Cognitive Behavioral Therapy for Adult Depression and Anxiety in Routine Secondary Care: Observational Study. J Med Internet Res. 2018 Nov 28;20(11):e10927. doi: 10.2196/10927. PMID 30487118
- [Background] Richards D, Richardson T. Computer-based psychological treatments for depression: a systematic review and meta-analysis. Clin Psychol Rev. 2012 Jun;32(4):329-42. doi: 10.1016/j.cpr.2012.02.004. Epub 2012 Feb 28. PMID 22466510
- [Background] Sasso KE, Strunk DR. Thin slice ratings of client characteristics in intake assessments: predicting symptom change and dropout in cognitive therapy for depression. Behav Res Ther. 2013 Aug;51(8):443-50. doi: 10.1016/j.brat.2013.04.007. Epub 2013 May 7. PMID 23747583
- [Background] Thase ME. The multifactorial presentation of depression in acute care. J Clin Psychiatry. 2013;74 Suppl 2:3-8. doi: 10.4088/JCP.12084su1c.01. PMID 24191971
- [Background] Titov N, Dear B, Nielssen O, Staples L, Hadjistavropoulos H, Nugent M, Adlam K, Nordgreen T, Bruvik KH, Hovland A, Repal A, Mathiasen K, Kraepelien M, Blom K, Svanborg C, Lindefors N, Kaldo V. ICBT in routine care: A descriptive analysis of successful clinics in five countries. Internet Interv. 2018 Jul 26;13:108-115. doi: 10.1016/j.invent.2018.07.006. eCollection 2018 Sep. PMID 30206525
- [Background] van Ballegooijen W, Cuijpers P, van Straten A, Karyotaki E, Andersson G, Smit JH, Riper H. Adherence to Internet-based and face-to-face cognitive behavioural therapy for depression: a meta-analysis. PLoS One. 2014 Jul 16;9(7):e100674. doi: 10.1371/journal.pone.0100674. eCollection 2014. PMID 25029507
- [Background] Setia S, Furtner D, Bendahmane M, Tichy M. Success4life Youth Empowerment for Promoting Well-being and Boosting Mental Health: Protocol for an Experimental Study. JMIR Res Protoc. 2022 Sep 14;11(9):e38463. doi: 10.2196/38463. PMID 36041997
- [Background] Vygotsky, L. S., & Cole, M. (1978). Mind in society: Development of higher psychological processes. Harvard University Press.
- [Background] Shafran R, Clark DM, Fairburn CG, Arntz A, Barlow DH, Ehlers A, Freeston M, Garety PA, Hollon SD, Ost LG, Salkovskis PM, Williams JM, Wilson GT. Mind the gap: Improving the dissemination of CBT. Behav Res Ther. 2009 Nov;47(11):902-9. doi: 10.1016/j.brat.2009.07.003. Epub 2009 Aug 6. PMID 19664756
- [Background] Kuyken W, Warren FC, Taylor RS, Whalley B, Crane C, Bondolfi G, Hayes R, Huijbers M, Ma H, Schweizer S, Segal Z, Speckens A, Teasdale JD, Van Heeringen K, Williams M, Byford S, Byng R, Dalgleish T. Efficacy of Mindfulness-Based Cognitive Therapy in Prevention of Depressive Relapse: An Individual Patient Data Meta-analysis From Randomized Trials. JAMA Psychiatry. 2016 Jun 1;73(6):565-74. doi: 10.1001/jamapsychiatry.2016.0076. PMID 27119968
- [Background] Rosendahl, H., Davidsen, M., Møller, S. R., Román, J. E. I., Kragelund, K., Christensen, A. I., & Ekholm, O. (2022). Danskernes sundhed: Den nationale sundhedsprofil 2021
- [Background] Reynolds CF 3rd, Cuijpers P, Patel V, Cohen A, Dias A, Chowdhary N, Okereke OI, Dew MA, Anderson SJ, Mazumdar S, Lotrich F, Albert SM. Early intervention to reduce the global health and economic burden of major depression in older adults. Annu Rev Public Health. 2012 Apr;33:123-35. doi: 10.1146/annurev-publhealth-031811-124544. PMID 22429161
- [Background] Pedersen MK, Mohammadi R, Mathiasen K, Elmose M. Internet-based cognitive behavioral therapy for anxiety in an outpatient specialized care setting: A qualitative study of the patients' experience of the therapy. Scand J Psychol. 2020 Dec;61(6):846-854. doi: 10.1111/sjop.12665. Epub 2020 Jul 23. PMID 32705703
- [Background] Mathiasen K, Andersen TE, Lichtenstein MB, Ehlers LH, Riper H, Kleiboer A, Roessler KK. The Clinical Effectiveness of Blended Cognitive Behavioral Therapy Compared With Face-to-Face Cognitive Behavioral Therapy for Adult Depression: Randomized Controlled Noninferiority Trial. J Med Internet Res. 2022 Sep 7;24(9):e36577. doi: 10.2196/36577. PMID 36069798
- [Background] Lutz W, Arndt A, Rubel J, Berger T, Schroder J, Spath C, Meyer B, Greiner W, Grafe V, Hautzinger M, Fuhr K, Rose M, Nolte S, Lowe B, Hohagen F, Klein JP, Moritz S. Defining and Predicting Patterns of Early Response in a Web-Based Intervention for Depression. J Med Internet Res. 2017 Jun 9;19(6):e206. doi: 10.2196/jmir.7367. PMID 28600278
- [Background] Laynard, R., Clark, D., Knapp, M., & Mayraz, G. (2007). Cost-benefit analysis of psychological therapy. National Institute Economic Review, 202(1), 90-98.
- [Background] Lawler K, Earley C, Timulak L, Enrique A, Richards D. Dropout From an Internet-Delivered Cognitive Behavioral Therapy Intervention for Adults With Depression and Anxiety: Qualitative Study. JMIR Form Res. 2021 Nov 12;5(11):e26221. doi: 10.2196/26221. PMID 34766909
- [Background] Kuyken W, Watkins E, Holden E, White K, Taylor RS, Byford S, Evans A, Radford S, Teasdale JD, Dalgleish T. How does mindfulness-based cognitive therapy work? Behav Res Ther. 2010 Nov;48(11):1105-12. doi: 10.1016/j.brat.2010.08.003. Epub 2010 Aug 13. PMID 20810101
- [Background] Klein T, Breilmann J, Schneider C, Girlanda F, Fiedler I, Dawson S, Crippa A, Priebe S, Barbui C, Becker T, Kosters M. Dose-response relationship in cognitive behavioral therapy for depression: A nonlinear metaregression analysis. J Consult Clin Psychol. 2024 May;92(5):296-309. doi: 10.1037/ccp0000879. PMID 38829329
- [Background] Karyotaki E, Efthimiou O, Miguel C, Bermpohl FMG, Furukawa TA, Cuijpers P; Individual Patient Data Meta-Analyses for Depression (IPDMA-DE) Collaboration; Riper H, Patel V, Mira A, Gemmil AW, Yeung AS, Lange A, Williams AD, Mackinnon A, Geraedts A, van Straten A, Meyer B, Bjorkelund C, Knaevelsrud C, Beevers CG, Botella C, Strunk DR, Mohr DC, Ebert DD, Kessler D, Richards D, Littlewood E, Forsell E, Feng F, Wang F, Andersson G, Hadjistavropoulos H, Christensen H, Ezawa ID, Choi I, Rosso IM, Klein JP, Shumake J, Garcia-Campayo J, Milgrom J, Smith J, Montero-Marin J, Newby JM, Breton-Lopez J, Schneider J, Vernmark K, Bucker L, Sheeber LB, Warmerdam L, Farrer L, Heinrich M, Huibers MJH, Kivi M, Kraepelien M, Forand NR, Pugh N, Lindefors N, Lintvedt O, Zagorscak P, Carlbring P, Phillips R, Johansson R, Kessler RC, Brabyn S, Perini S, Rauch SL, Gilbody S, Moritz S, Berger T, Pop V, Kaldo V, Spek V, Forsell Y. Internet-Based Cognitive Behavioral Therapy for Depression: A Systematic Review and Individual Patient Data Network Meta-analysis. JAMA Psychiatry. 2021 Apr 1;78(4):361-371. doi: 10.1001/jamapsychiatry.2020.4364. PMID 33471111
- [Background] Karyotaki E, Kemmeren L, Riper H, Twisk J, Hoogendoorn A, Kleiboer A, Mira A, Mackinnon A, Meyer B, Botella C, Littlewood E, Andersson G, Christensen H, Klein JP, Schroder J, Breton-Lopez J, Scheider J, Griffiths K, Farrer L, Huibers MJH, Phillips R, Gilbody S, Moritz S, Berger T, Pop V, Spek V, Cuijpers P. Is self-guided internet-based cognitive behavioural therapy (iCBT) harmful? An individual participant data meta-analysis. Psychol Med. 2018 Nov;48(15):2456-2466. doi: 10.1017/S0033291718000648. Epub 2018 Mar 15. PMID 29540243
- [Background] Karyotaki E, Riper H, Twisk J, Hoogendoorn A, Kleiboer A, Mira A, Mackinnon A, Meyer B, Botella C, Littlewood E, Andersson G, Christensen H, Klein JP, Schroder J, Breton-Lopez J, Scheider J, Griffiths K, Farrer L, Huibers MJ, Phillips R, Gilbody S, Moritz S, Berger T, Pop V, Spek V, Cuijpers P. Efficacy of Self-guided Internet-Based Cognitive Behavioral Therapy in the Treatment of Depressive Symptoms: A Meta-analysis of Individual Participant Data. JAMA Psychiatry. 2017 Apr 1;74(4):351-359. doi: 10.1001/jamapsychiatry.2017.0044. PMID 28241179
- [Background] Karyotaki E, Kleiboer A, Smit F, Turner DT, Pastor AM, Andersson G, Berger T, Botella C, Breton JM, Carlbring P, Christensen H, de Graaf E, Griffiths K, Donker T, Farrer L, Huibers MJ, Lenndin J, Mackinnon A, Meyer B, Moritz S, Riper H, Spek V, Vernmark K, Cuijpers P. Predictors of treatment dropout in self-guided web-based interventions for depression: an 'individual patient data' meta-analysis. Psychol Med. 2015 Oct;45(13):2717-26. doi: 10.1017/S0033291715000665. Epub 2015 Apr 17. PMID 25881626
- [Background] Hayes, S. C., Strosahl, K. D., & Wilson, K. G. (1999). Acceptance and commitment therapy (Vol. 6). Guilford Press
- [Background] Gilbert P. The origins and nature of compassion focused therapy. Br J Clin Psychol. 2014 Mar;53(1):6-41. doi: 10.1111/bjc.12043. PMID 24588760
- [Background] Cuijpers P, Noma H, Karyotaki E, Vinkers CH, Cipriani A, Furukawa TA. A network meta-analysis of the effects of psychotherapies, pharmacotherapies and their combination in the treatment of adult depression. World Psychiatry. 2020 Feb;19(1):92-107. doi: 10.1002/wps.20701. PMID 31922679
- [Background] Chand SP, Kuckel DP, Huecker MR. Cognitive Behavior Therapy. 2023 May 23. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470241/ PMID 29261869
- [Background] Butler AC, Chapman JE, Forman EM, Beck AT. The empirical status of cognitive-behavioral therapy: a review of meta-analyses. Clin Psychol Rev. 2006 Jan;26(1):17-31. doi: 10.1016/j.cpr.2005.07.003. Epub 2005 Sep 30. PMID 16199119
- [Background] Bliss, J., Askew, M., & Macrae, S. (1996). Effective teaching and learning: Scaffolding revisited. Oxford Review of Education, 22(1), 37-61.
- [Background] Beck, J. S. (2020). Cognitive behavior therapy: Basics and beyond (3rd ed.). Guilford Publications.
- [Background] Beck, A. T. (1979). Cognitive therapy of depression. Guilford Press.
- [Background] Barrett MS, Chua WJ, Crits-Christoph P, Gibbons MB, Casiano D, Thompson D. EARLY WITHDRAWAL FROM MENTAL HEALTH TREATMENT: IMPLICATIONS FOR PSYCHOTHERAPY PRACTICE. Psychotherapy (Chic). 2008 Jun 1;45(2):247-267. doi: 10.1037/0033-3204.45.2.247. PMID 19838318
- [Background] Barak, A., Hen, L., Boniel-Nissim, M., & Shapira, N. A. (2008). A comprehensive review and a meta-analysis of the effectiveness of internet-based psychotherapeutic interventions. Journal of Technology in Human Services, 26(2-4), 109-160
- [Background] Andrews G, Basu A, Cuijpers P, Craske MG, McEvoy P, English CL, Newby JM. Computer therapy for the anxiety and depression disorders is effective, acceptable and practical health care: An updated meta-analysis. J Anxiety Disord. 2018 Apr;55:70-78. doi: 10.1016/j.janxdis.2018.01.001. Epub 2018 Feb 1. PMID 29422409
- [Background] Alonso J, Codony M, Kovess V, Angermeyer MC, Katz SJ, Haro JM, De Girolamo G, De Graaf R, Demyttenaere K, Vilagut G, Almansa J, Lepine JP, Brugha TS. Population level of unmet need for mental healthcare in Europe. Br J Psychiatry. 2007 Apr;190:299-306. doi: 10.1192/bjp.bp.106.022004. PMID 17401035
- [Background] Alonso J, Angermeyer MC, Bernert S, Bruffaerts R, Brugha TS, Bryson H, de Girolamo G, Graaf R, Demyttenaere K, Gasquet I, Haro JM, Katz SJ, Kessler RC, Kovess V, Lepine JP, Ormel J, Polidori G, Russo LJ, Vilagut G, Almansa J, Arbabzadeh-Bouchez S, Autonell J, Bernal M, Buist-Bouwman MA, Codony M, Domingo-Salvany A, Ferrer M, Joo SS, Martinez-Alonso M, Matschinger H, Mazzi F, Morgan Z, Morosini P, Palacin C, Romera B, Taub N, Vollebergh WA; ESEMeD/MHEDEA 2000 Investigators, European Study of the Epidemiology of Mental Disorders (ESEMeD) Project. Prevalence of mental disorders in Europe: results from the European Study of the Epidemiology of Mental Disorders (ESEMeD) project. Acta Psychiatr Scand Suppl. 2004;(420):21-7. doi: 10.1111/j.1600-0047.2004.00327.x. PMID 15128384
- See also: The home page of the PERSONAE project — https://personae.cedip.dk/